CLINICAL TRIAL: NCT06384040
Title: Immuno-based Profiling of knEe OA Patients to Predict reSponse to Regenerative Treatment
Acronym: IMPRESA
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: GR-2019-12370692
Record Dates: First submitted 2024-04-05; First posted 2024-04-25 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRP responder: response to treatment will be established in the presence of >40% improvement of pain and/or motility
  Interventions: Procedure: platelet-rich plasma knee injection
- PRP non responder: response to treatment will be established in the presence of <40% improvement of pain and/or motility
  Interventions: Procedure: platelet-rich plasma knee injection

INTERVENTIONS:
Procedure: platelet-rich plasma knee injection — platelet-rich plasma knee injection and observation for 12 months for definition of responder and non responder

SUMMARY:
Osteoarthritis (OA) is a highly prevalent degenerative musculoskeletal disease and a major cause of chronic disability worldwide. Its multifactorial origin contributes to determine the heterogeneous phenotypes and one unmet need is the lack of biomarkers to predict the individual response. Platelet-rich-plasma (PRP) injection is a minimally invasive autologous blood-derived approach for which we plan to define specific knee profiles predictive of response. We will take advantage of a unique multidisciplinary approach aimed at analysing clinics, imaging, and biomarkers of associated with clinical response. We will focus on inflammatory (Wnt system, IL1 pathway, PTX3) and antioxidant (primarily, DPP3/Keap1/Nrf2) pathways. We foresee that our results will allow a better allocation of immunomodulatory and regenerative therapies for a personalized approach in knee OA thus maximising the effectiveness of the healthcare allocation.

ELIGIBILITY:
Inclusion Criteria:

* men/women, aged >40 - <75 years), OA grade 2-3, BMI <40, baseline WOMAC PAIN >1.75 -<4, >1 conservative therapy failed. Diagnosis of knee OA according to the American College of Rheumatology (ACR) classification criteria (Altman, 1986) .
* Ability to give informed consent.

Exclusion Criteria:

* Presence of active infection or abnormal knee effusion on Day 1 at pre-injection of PRP
* Diagnosis of chronic inflammatory disease (i.e. rheumatoid arthritis, reactive arthritis, psoriatic arthritis, chondromalacia, arthritis secondary to other inflammatory diseases)
* Untreated acute traumatic injury, presence of a symptomatic meniscal tear, valgus/varus deformity judged by the investigator to be clinically significant, in the index knee
* Recent (within 3-6 months) arthroscopy, open surgery, intra-articular steroid injections, intra-articular hyaluronic acid (HA) injections, systemic steroid treatment, malignancy
* Any serious, non-malignant, significant, acute, or chronic medical condition or active psychiatric illness that, in the investigator's opinion, could compromise patient safety, limit the patient's ability to complete the study, and/or compromise the objectives of the study.
* Recent (within 30 days) use of any investigational drug or device prior to screening

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Knee OA patients will be enrolled at the outpatient clinic of UO1 and UO2 during the routine activity. They will receive a thorough description of the project and, if willing to participate, they will sign the informed consent. The patient number needed in the study has been calculated to ensure a proper representation of the described phenotypes (Soul J et al, 2018). The patients will undergo imaging and clinical evaluations; the respective results will be analysed and correlated with laboratory evaluations. Moreover, all patients will undergo biologic sample harvesting (as detailed below) and afterwards PRP injection. We will collect peripheral blood (PB) samples and, when available, synovial fluid (SF) from the patients prior to PRP injection
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
knee OA patients focusing on changes in Wnt and IL1-ß signalling and PTX3 expression | 18 months
  We will collect peripheral blood (PB) samples and cellular and molecular components in these samples will be characterized by measuring gene expression and protein levels of soluble factors involved in inflammatory pathways, with specific attention to Wnt and IL1 signaling pathways, and PTX3, and by performing a complete immunophenotype. We will use computational clustering approaches applied to single cell FACS data (Phenograph, FlowSOM, or similar) to identify phenotypic subsets in an unbiased way.

SECONDARY OUTCOMES:
To assess the overall oxidative status and antioxidant capacity of the enrolled OA patients and its possible prognostic role with respect to response to PRP treatment | 36 months
  We will define the overall oxidative status in the patients at baseline, by measuring a set of parameters related to enzymatic and non-enzymatic antioxidant systems, comprising the total antioxidant capacity, total glutathione, catalase activity, advanced glycation end products, HNE adducts, vitamin E and C, in the serum and SF, when available.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided